CLINICAL TRIAL: NCT02788695
Title: The Northern Ireland Sensory Ageing Study
Acronym: NISA
Status: Completed | Type: Observational
Sponsor: Queen's University, Belfast (Other)
Collaborators: College of Optometrists (Unknown)
Responsible Party: Principal Investigator, Ruth Hogg, Doctor, Queen's University, Belfast
Other Study IDs: 14.25
Record Dates: First submitted 2016-04-28; First posted 2016-06-02 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Aging
Keywords: Visual Nonspecific

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1 - aged 20-90 years: 25 participants from each decade from 20-90. Those from 50+ will be recruited from the NICOLA study and retinal/lens images assessed to confirm normality.
- Group 2: aged 60 years: Group 2: 250 participants NICOLA participants aged 60 will be invited to participate; only those whose ocular images confirm normality will be included.

SUMMARY:
A visual function focused add-on study to the Northern Ireland Cohort for the Longitudinal Study of Ageing (NICOLA). There are three key aims:

1. Quantify age-related decline in a variety of visual functions within a populations based cohort.
2. Explore the mechanisms underlying age-related visual impairments.
3. Investigate how visual function impacts vision related quality of life.

DETAILED DESCRIPTION:
The investigators propose to put together a battery of test to assess different aspects of visual function and apply them to two groups of participants in order to explore differences in chronological and physiological aging.

Group 1: 25 participants from each decade from 20-90. Those from 50+ will be recruited from the NICOLA study and retinal/lens images assessed to confirm normality (drusen <63µm or clear retina, LOCS III <1). Those younger will be recruited via advertisements in the University and targeting friends and relatives or NICOLA participants. This will enable the rate of decline with age to be calculated. Linear, bilinear, and simple nonlinear candidate functions of parameter vs. age will be applied to determine which best characterises the change.

Group 2: 250 participants NICOLA participants aged 60 will be invited to participate; only those whose ocular images confirm normality will be included. This will enable mechanisms underlying individual differences in aging to be investigated. Normal aging will be determined from group 1 analysis and participants will be able to be categorised as aging well or aging poorly. Multivariate regression analysis will be used to investigate the relationship between visual function and lifestyle and environmental factors. Principal components analysis will be used to look at the relationships between visual parameters. These participants will also be asked to complete the NEIVFQ-25, to characterise visual function related quality of life and this will be compared with their measured visual function.

Visual function parameters measured after protocol refraction will include: Photopic and mesopic visual acuity and contrast sensitivity using City Occupational acuity-plus software17, near visual acuity, reading speed and SKILL card18, MAIA microperimetry and cone dark adaptation.19 Intra-ocular scatter will be assessed using the Oculus C-quant to assess the extent to which ocular factors are degrading vision.20 Three-point vernier acuity will also be measured as this is thought to stay stable throughout life.15 Time will be taken to ensure participants receive sufficient training to produce reliable thresholds.

All study visits will occur at the Welcome-Wolfson Clinic Research Facility.

ELIGIBILITY:
Inclusion Criteria:

* No diagnosed ocular disease.
* Non-diabetic.

Exclusion Criteria:

* Any diagnosed ocular disease.
* Diabetic.
* Cognitive impairment.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 25 participants from each decade from 20-90. Those from 50+ will be recruited from the NICOLA study. 250 participants NICOLA participants aged 60 will be invited to participate; only those whose ocular images confirm normality will be included.
Sampling Method: Probability Sample
Enrollment: 842 (Actual)
Dates: Start 2014-11; Primary Completion 2018-04-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of decline of visual function with age | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Hogg, Principal Investigator — Queen's University, Belfast
Locations (1):
- NI Clinical Research Facility, Belfast, Northern Ireland, United Kingdom

IPD SHARING:
Plan to Share IPD: No